CLINICAL TRIAL: NCT02266498
Title: Single-dose Pharmacokinetics of 2.5 mg BIBB 515 BS and Effect of Food After Oral Administration of Capsules to Healthy Subjects (Randomized, 2-way-cross-over, Open Study)
Brief Title: Pharmacokinetics of BIBB 515 BS and Effect of Food After Oral Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 525.4
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — CD36 Antigens

ARMS (2):
- BIBB 515 BS after a standard breakfast (Experimental)
  Interventions: Drug: BIBB 515 BS; Other: Standard breakfast (40 g fat)
- BIBB 515 BS (Active Comparator)
  Interventions: Drug: BIBB 515 BS

INTERVENTIONS:
Drug: BIBB 515 BS
Other: Standard breakfast (40 g fat)
  Arms: BIBB 515 BS after a standard breakfast

SUMMARY:
To assess the effect of a breakfast (40 g fat) on single dose pharmacokinetics of a 2.5 mg BIBB 515 dose in capsules as well as the tolerability of BIBB 515 BS capsules

ELIGIBILITY:
Inclusion Criteria:

* Healthy male caucasian subjects as determined by results of screening
* Written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurologic disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (≤ 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation > 100 ml (≤ 4 weeks prior to administration or during the trial)
* Excessive physical activities (≤ 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1998-06; Primary Completion 1998-07 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | Up to 48 hours after drug administration
Time to reach maximum concentration of the analyte in plasma (tmax) | Up to 48 hours after drug administration
Apparent terminal elimination half-life of the analyte in plasma (t1/2) | Up to 48 hours after drug administration
Area under the concentration-time curve of the analyte in plasma at different time points (AUC) | Up to 48 hours after drug administration
Total mean residence time of the analyte in the body (MRTtot) | Up to 48 hours after drug administration
Apparent clearance of the analyte in plasma after extravascular multiple dose administration (CL/f) | Up to 48 hours after drug administration
Apparent volume of distribution of the analyte during the terminal phase (Vz/f) | Up to 48 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | Up to 48 hours after drug administration
Number of patients with adverse events | Up to 48 hours after last drug administration
Global clinical assessment by the investigator | Day 3 after last drug administration